CLINICAL TRIAL: NCT04628754
Title: A Randomized Control Trial of a Primary Care Intervention to Reverse Frailty and Enhance Resilience Through Resistance Exercise and Dietary Protein Education (REFEREE) Among Community Dwelling Adults Aged 65 and Over
Brief Title: A Randomized Control Trial of an Intervention to Reverse Frailty and Enhance Resilience Through Exercise and Education
Acronym: REFEREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, John Travers, Doctor, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REFEREE
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Frailty; Sarcopenia
Keywords: Resilience; Primary-care; Intervention; Exercise; Protein; Diet; Community
MeSH Terms: conditions — Frailty; Sarcopenia; Motor Activity | interventions — Exercise; Proteins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Resistance exercise and dietary protein guidance
  Interventions: Other: Exercise and protein
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Exercise and protein — Home based exercise regime and dietary protein guidance
  Arms: Intervention

SUMMARY:
Resistance training done at home and protein supplementation may be the most effective and easiest to implement interventions to reverse frailty and build resilience. However, it is not common practice to offer and support such interventions in primary care.

This study provides an opportunity to assess the effectiveness of an optimised intervention with community-dwelling adults aged 65 and over, whose baseline clinical frailty score is not worse than mild (i.e. 5 or less), evaluate improvements in health outcomes and demonstrate how the intervention may be incorporated efficiently in clinical practice. The results are intended to encourage mainstream adoption of practical interventions to reverse clinical frailty and build resilience in primary care.

An intervention with ten recommended resistance exercises and dietary guidance on protein consumption has been derived from findings of our systematic review and meta-analysis and optimised through a patient and public involvement (PPI) process and feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or older at baseline
* Rockwood clinical frailty scale score 4 or 5 (vulnerable or mildly frail)
* Able and willing to provide informed consent and to comply with the requirements of this study protocol

Exclusion Criteria:

* Rockwood clinical frailty scale score > 5
* End of life care
* Persons in residential care home
* Concurrent malignancy CKD stage 3 or 4
* Coded diagnosis of severe dementia as per GP or consultant geriatrician diagnosis or baseline Montreal Cognitive assessment (MoCA) score <= 10
* Persons unable to engage in discussion on frailty due to acute care needs or determined to be inappropriate by GP (e.g., needing transfer to ED or acutely unwell or disorders resulting in intolerance of the intervention)
* Subjects unable to provide written informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 169 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Frailty status | 3 months
  Frailty status as measured by SHARE-frailty instrument measurement

SECONDARY OUTCOMES:
Clinical frailty status | 3 months
  Clinical frailty status measured by Clinical Frailty Scale 1 to 9, 9 is worse
Sarcopenia/ muscle mass | 3 months
  Sarcopenia/ muscle mass measured by bioelectrical impedance
Ease of the intervention | 3 months
  Ease of the intervention measured on a five-point scale: 'very easy', 'somewhat easy', 'neither easy nor hard', 'somewhat hard', or 'very hard'
Subjective difference to general health | 3 months
  Difference to general health as a result of the exercises measured on a five-point scale: 'much better', 'slightly better', 'about the same', 'slightly worse' or 'much worse'
Bone mass | 3 months
  Bone mass measured by bioelectrical impedance
Body fat | 3 months
  measured by bioelectrical impedance
Biological age | 3 months
  measured by bioelectrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Marie Therese Cooney, PhD, Study Director — University College Dublin
Locations (1):
- Beechlawn Medical Centre, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Travers J, Romero-Ortuno R, Power D, Doran P, Langan J, MacNamara F, McCormack D, McDermott C, McEntire J, McKiernan J, Vencken S, Murphy AW, Murphy PJ, Ni She E, O'Shea D, Cooney MT. Protocol for a randomised controlled trial of a primary care intervention to Reverse Frailty and Enhance Resilience through Exercise and dietary protein Education (REFEREE) in community-dwelling adults aged 65 and over. HRB Open Res. 2021 Apr 21;3:91. doi: 10.12688/hrbopenres.13188.2. eCollection 2020. PMID 33977224
- See also: Published protocol for this trial — https://hrbopenresearch.org/articles/3-91